CLINICAL TRIAL: NCT02540096
Title: Effects of Mental Practice for Mobility in Post-stroke Hemiparesis: Randomized Controlled Trial of Efficacy.
Brief Title: Effects of Mental Practice for Mobility in Post-stroke Hemiparesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Zaqueline F. Guerra, MSc, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43659515.4.0000.5103
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Stroke; Hemiparesis
Keywords: mental practice; motor imagery; hemiparesis; stroke; gait; mobility
MeSH Terms: conditions — Stroke; Paresis | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Mental Practice) (Experimental): Participants will be submitted to individual and structured physiotherapy sessions (the same as the control groups). They will also participate in a structured mental practice session (lasting 30 minutes and three times a week), totaling 12 sessions at the end of this intervention.
  Interventions: Other: Mental practice
- Control group (Placebo Comparator): Participants will be submitted to individual and structured physiotherapy sessions lasting 40 minutes. They will also participate in a cognitive training and relaxation session (lasting 30 minutes, three times a week), totaling 12 sessions.
  Interventions: Other: Cognitive training and Relaxation

INTERVENTIONS:
Other: Mental practice — The sessions will be individualized and carried out in a peaceful setting.The aim of the mental practice protocol was to promote motor imagery of the following activities: get up from a chair and walk and sit, which enrolls the basic and instrumental activities of daily living. The sessions will consist of six steps: (1) "Physical Practice" (2) "Familiarization" (3) "Memory" (4) "Relaxation" (5) "Repeat" and (6) "post-practice mental relaxation". After the mental practice session, participants will be submitted to individual and structured physiotherapy sessions (the same as the control groups).
  Arms: Intervention (Mental Practice)
Other: Cognitive training and Relaxation — Cognitive training and relaxation session (lasting 30 minutes, three times a week), totaling 12 sessions. The sessions will consist of calculations, memorization, imagination and body relaxation exercises. These sessions will not have any motor imagery. After the cognitive training and relaxation session, participants will be submitted to individual and structured physiotherapy sessions lasting 40 minutes with muscle strengthening and stretching exercises.
  Arms: Control group

SUMMARY:
Stroke is a neurovascular event characterized by impaired blood supply to the brain due to rupture or obstruction of certain cerebral arteries, which often results in hemiparesis and can affect individuals of any age and sex, being prevalent in the elderly population.

Among the main treatments available for stroke rehabilitation, most of them demands an appropriate structure and high-qualified personnel. Searching for more affordable treatment options, several studies suggest the use of mental practice with motor imagery as a potential therapeutic tool, since it can be performed at any place or any time the patient wishes, including their own homes.

Motor imagery can be defined as the covert cognitive process of imagining a movement of your own body(-part) without actually moving that body(-part).

Within this context, the objective of this study is to investigate the effects of mental practice for mobility, gait function and speed and muscle strength of the lower limb in subacute post-stroke hemiparesis.

DETAILED DESCRIPTION:
Post-stroke patients will be invited to participate after hospital discharge, based on inclusion and exclusion criteria. Then, after acceptance, participants will be randomized (block strategy) into two groups: Control group (Physiotherapy and Cognitive mental exercise) and Intervention group (Physiotherapy and Mental Practice group).

At baseline, 4 weeks (end of intervention) and 6 weeks, participants will be evaluated through the following tests: Timed-Up and Go test, 5-Meter Walk Test, TUG-ABS, WHOQOL-Bref, DASS-21 and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* hemiparesis after ischemic stroke (15 to 180 days after the event);
* only one cerebral hemisphere affected;
* no chemical, alcohol or drug dependency;
* Score average ≥ 2,5 point in the instrument "Visual and Kinesthetic Imagery Questionnaire" (KIVQ-10);
* No cognitive impairment (18 points in the Mini-Mental State Examination - 0-4 years of educations and 24 points (>4 years of education);
* Not participating in any other type of physiotherapy or physical activity during the study period;
* Complaining of difficulty in gait and mobility after stroke;
* Able to stand up from a chair and walk some distance with or without auxiliary device;

Exclusion Criteria:

* Hemorrhagic or ischemic progressing to hemorrhagic stroke;
* Score ≥ 4 on the Visual Analogue Pain Scale;
* Score ≥ 2 on the modificator Ashworth scale;
* Visual disabilities;
* Severe Aphasia;
* Cardiovascular instability and/or other neurological disorders that may impair the mobility and gait.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-01 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in Timed Up and Go (TUG) | 1 week before intervention; 4 weeks after intervention; 6 weeks after intervention
  This is a measure that examines the participant's basic mobility skills by measuring seconds to rise from sitting, walk 3 meters, return, and sitting down
5-Meter Walk Test | 1 week before intervention; 4 weeks after intervention; 6 weeks after intervention
  This is a measure that examines the participant's gait speed (cut off 6 seconds)

SECONDARY OUTCOMES:
Change in Muscle strength | 1 week before intervention; 4 weeks after intervention; 6 weeks after intervention
  Hand-held dynamometer (HDD) for measuring lower-limb muscle strength
Change in Quality of life | 1 week before intervention; 4 weeks after intervention; 6 weeks after intervention
  Using World Health Organization Quality of Life Instrument (WHOQOL-Bref)
Change in Mental health | 1 week before intervention; 4 weeks after intervention; 6 weeks after intervention
  Using Depression, anxiety and stress scale (DASS-21)
Change in TUG-ABS | 1 week before intervention; 4 weeks after intervention; 6 weeks after intervention
  The Timed "Up and Go" Assessment of Biomechanical Strategies (TUG-ABS)

CONTACTS AND LOCATIONS:
Overall Officials: Zaqueline F Guerra, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- Zaqueline Fernandes Guerra, Juiz de Fora, Brazil

REFERENCES:
- [Background] Paolucci S, Antonucci G, Grasso MG, Morelli D, Troisi E, Coiro P, Bragoni M. Early versus delayed inpatient stroke rehabilitation: a matched comparison conducted in Italy. Arch Phys Med Rehabil. 2000 Jun;81(6):695-700. doi: 10.1016/s0003-9993(00)90095-9. PMID 10857508
- [Background] Hadidi N, Buckwalter K, Lindquist R, Rangen C. Lessons learned in recruitment and retention of stroke survivors. J Neurosci Nurs. 2012 Apr;44(2):105-10. doi: 10.1097/JNN.0b013e3182478c96. PMID 22367274
- [Background] Zhang S, He WB, Chen NH. Causes of death among persons who survive an acute ischemic stroke. Curr Neurol Neurosci Rep. 2014 Aug;14(8):467. doi: 10.1007/s11910-014-0467-3. PMID 24951970
- [Background] Page SJ, Dunning K, Hermann V, Leonard A, Levine P. Longer versus shorter mental practice sessions for affected upper extremity movement after stroke: a randomized controlled trial. Clin Rehabil. 2011 Jul;25(7):627-37. doi: 10.1177/0269215510395793. Epub 2011 Mar 22. PMID 21427151
- [Background] Page SJ. Mental practice: a promising restorative technique in stroke rehabilitation. Top Stroke Rehabil. 2001 Autumn;8(3):54-63. doi: 10.1310/7WDU-2P4U-V2EA-76F8. PMID 14523738
- [Background] Page SJ, Levine P, Leonard AC. Effects of mental practice on affected limb use and function in chronic stroke. Arch Phys Med Rehabil. 2005 Mar;86(3):399-402. doi: 10.1016/j.apmr.2004.10.002. PMID 15759218
- [Background] Lotze M, Cohen LG. Volition and imagery in neurorehabilitation. Cogn Behav Neurol. 2006 Sep;19(3):135-40. doi: 10.1097/01.wnn.0000209875.56060.06. PMID 16957491
- [Background] Sirigu A, Duhamel JR. Motor and visual imagery as two complementary but neurally dissociable mental processes. J Cogn Neurosci. 2001 Oct 1;13(7):910-9. doi: 10.1162/089892901753165827. PMID 11595094
- [Background] Jeannerod M. Neural simulation of action: a unifying mechanism for motor cognition. Neuroimage. 2001 Jul;14(1 Pt 2):S103-9. doi: 10.1006/nimg.2001.0832. PMID 11373140
- [Background] Malouin F, Richards CL, Jackson PL, Lafleur MF, Durand A, Doyon J. The Kinesthetic and Visual Imagery Questionnaire (KVIQ) for assessing motor imagery in persons with physical disabilities: a reliability and construct validity study. J Neurol Phys Ther. 2007 Mar;31(1):20-9. doi: 10.1097/01.npt.0000260567.24122.64. PMID 17419886
- [Background] Malouin F, Richards CL, Doyon J, Desrosiers J, Belleville S. Training mobility tasks after stroke with combined mental and physical practice: a feasibility study. Neurorehabil Neural Repair. 2004 Jun;18(2):66-75. doi: 10.1177/0888439004266304. PMID 15228801
- [Background] Malouin F, Richards CL, Durand A, Doyon J. Added value of mental practice combined with a small amount of physical practice on the relearning of rising and sitting post-stroke: a pilot study. J Neurol Phys Ther. 2009 Dec;33(4):195-202. doi: 10.1097/NPT.0b013e3181c2112b. PMID 20208464
- [Background] Malouin F, Richards CL, Durand A, Doyon J. Clinical assessment of motor imagery after stroke. Neurorehabil Neural Repair. 2008 Jul-Aug;22(4):330-40. doi: 10.1177/1545968307313499. Epub 2008 Mar 6. PMID 18326057
- [Background] Hesse S, Schauer M, Malezic M, Jahnke M, Mauritz KH. Quantitative analysis of rising from a chair in healthy and hemiparetic subjects. Scand J Rehabil Med. 1994 Sep;26(3):161-6. PMID 7801066
- [Background] Decety J. The neurophysiological basis of motor imagery. Behav Brain Res. 1996 May;77(1-2):45-52. doi: 10.1016/0166-4328(95)00225-1. PMID 8762158
- [Background] Dunsky A, Dickstein R, Marcovitz E, Levy S, Deutsch JE. Home-based motor imagery training for gait rehabilitation of people with chronic poststroke hemiparesis. Arch Phys Med Rehabil. 2008 Aug;89(8):1580-8. doi: 10.1016/j.apmr.2007.12.039. PMID 18674992
- [Background] Braun S, Kleynen M, van Heel T, Kruithof N, Wade D, Beurskens A. The effects of mental practice in neurological rehabilitation; a systematic review and meta-analysis. Front Hum Neurosci. 2013 Aug 2;7:390. doi: 10.3389/fnhum.2013.00390. eCollection 2013. PMID 23935572
- [Background] Ietswaart M, Johnston M, Dijkerman HC, Joice S, Scott CL, MacWalter RS, Hamilton SJ. Mental practice with motor imagery in stroke recovery: randomized controlled trial of efficacy. Brain. 2011 May;134(Pt 5):1373-86. doi: 10.1093/brain/awr077. Epub 2011 Apr 22. PMID 21515905
- [Derived] Guerra ZF, Bellose LC, Ferreira AP, Faria CDCM, Paz CCSC, Lucchetti G. Effects of mental practice on mobility of individuals in the early subacute post-stroke phase: A randomized controlled clinical trial. J Bodyw Mov Ther. 2022 Oct;32:82-90. doi: 10.1016/j.jbmt.2022.04.018. Epub 2022 Apr 27. PMID 36180164